CLINICAL TRIAL: NCT07011030
Title: Comparison of the Use of a Bioimpedance Meter With Integretaed Electrodes and Osteodensitometry for the Diagnosis os Sarcopenia in the Elderly
Brief Title: Diagnosis of Sarcopenia in Older Adults
Acronym: SARCO-BIODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-PP-04
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
Keywords: sarcopenia; elderly; bioimpedance analysis; osteodensitometry
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skeletal muscle mass measurement (Experimental): Patients will undergo a:
  * Bioimpedance analysis with the Biody XpertZM 3 (bioimpedance device with integrated electrodes )
  * Osteodensitometer analysis with the SRATOS DR
  Interventions: Other: Measure of skeletal muscle mass

INTERVENTIONS:
Other: Measure of skeletal muscle mass — Bioimpedance analysis with integrated electrodes and osteodensitometry examination

SUMMARY:
Sarcopenia is defined as the loss of muscle strength and mass associated with aging and is one of the main causes of frailty in older people, and therefore of their ability to age gracefully. Given the aging of the French population, the diagnosis and management of this condition is a major public health issue and, in this context, it is therefore necessary to be able to quickly assess people's skeletal muscle mass.

In its recommendations, French National Authority for Health recommends the use osteodensitometry and bioimpedance analysis (BIA) to assess skeletal muscle mass in the limbs for the purpose of diagnosing sarcopenia. Traditionally, BIA assessment is performed while lying down using adhesive electrodes placed on the hands and feet. The Biody XpertZM3 is a BIA device that allows seated measurement using integrated electrodes, enabling skeletal muscle mass to be assessed by bioimpedance analysis without the use of adhesive electrodes. However, the measurement position could alter the impedances measured and therefore the results obtained compared to other devices on the market as well as osteodensitometer

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 60 or over already receiving care at the Day Hospital of the Rehabilitation, Independence and Aging Center or the Frailty Platform of the Rehabilitation, Independence and Aging Center.
* Patients affiliated with or covered by a social security system.
* Patients who have signed an informed consent form in advance.

Exclusion Criteria:

* Vulnerable persons as defined in Articles L1121-5 to -8
* People with pacemakers, implantable defibrillators, or other electronic medical devices
* Musculoskeletal disorders that prevent bioimpedance measurement in a seated position
* Any condition of fluid retention or dehydration
* Absence of a measurement site (muscle resection or amputation)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-09-23 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass | day 0
  Comparison of skeletal muscle mass of the limbs (in kg) obtained by bioimpedance analysis using integrated electrodes and using osteodensitometry

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric CHORIN, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France